CLINICAL TRIAL: NCT03077581
Title: The Efficacy of Three Different Surgically Infiltrated Local Anesthetic Techniques in Abdominoplasty
Brief Title: Comparison of Three Techniques for Analgesia After Abdominoplasty
Acronym: Maha1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, AlRefaey Kandeel, lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: D.Maha abdominoplasty
Record Dates: First submitted 2017-03-03; First posted 2017-03-13 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Abdominoplasty Patients

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transevrsus abdominus plane block group (Active Comparator)
  Interventions: Drug: Transevrsus abdominus plane block
- Rectus sheath block group (Active Comparator)
  Interventions: Drug: Rectus sheath block
- local infiltration group (Active Comparator)
  Interventions: Drug: local anesthesia infiltartion

INTERVENTIONS:
Drug: Transevrsus abdominus plane block — a blunt needle was advanced in the midaxillary line to reach the fascial layer between the internal oblique and transverse abdominis muscles detected by facial click sensation. The LA was slowly injected so as to detect any sign of toxicity or incorrect needle tip position (as resistance) requiring needle repositioning then TAPB was repeated on the opposite side.
  Arms: Transevrsus abdominus plane block group
Drug: Rectus sheath block — In RSB group, 2-3 cm from midline, about 3-5 cm above the umbilicus, the needle was advanced at right angle to the skin. The needle reaches the space between the posterior layer of the rectus sheath and rectus abdominis muscle detected by firm resistance of the posterior wall, The LA was slowly injected then the same steps were repeated on the other side.
  Arms: Rectus sheath block group
Drug: local anesthesia infiltartion — 40 mls of 0.255 bupivacaine will be infiltrated at skin incision
  Arms: local infiltration group

SUMMARY:
This study was conducted to demonstrate post-abdominoplasty analgesic duration consequent to three different surgically infiltrated LA techniques; bilateral TAPB, bilateral RSB and subcutaneous infiltration using the same volume of 0.25% bupivacaine (40 ml). Pain score, total analgesic rescue requests and the total amount of systemic rescue analgesia used in the first postoperative day in addition to any detected postoperative complications were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* all patients listed for abdominoplasty

Exclusion Criteria:

* allergy to bupivacaine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-06-05 (Estimated); Study Completion 2017-06-15 (Estimated)

PRIMARY OUTCOMES:
morphine consumption (mg) | up to 24 hours
  postoperative morphine consumption in milligrams in the 1st 24 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided